CLINICAL TRIAL: NCT06852664
Title: Improving Activity in Individuals With Cerebral Palsy
Acronym: Fitbit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Father Flanagan's Boys' Home (Other)
Responsible Party: Principal Investigator, Max Kurz, Director of PoWER Lab, Father Flanagan's Boys' Home
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-23-XP
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Fitbit; Mobility; Steps
MeSH Terms: conditions — Cerebral Palsy | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Cerebral Palsy participants will undergo baseline mobility/brain imaging/cognitive testing, receive motivational interviewing, and then repeat mobility/brain imaging testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cerebral Palsy Youth/Young Adults (Experimental): Baseline and 8-week assessments as well as 8 weeks of motivational interviewing 3x/week
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — The participants will meet with the research staff three times a week during the eight weeks of wearing the activity monitor via video or Webex call with a duration ideally not exceeding one hour. All staff involved in these coaching sessions have been MINT trained and certified and have mastered the skills of motivational interviewing. Their goal will be to discuss with the participant about how successful they have been or not been in increasing their daily step count and movement and discussing the barriers preventing them from achieving that goal. Open-ended questions, affirmations, reflections, summaries, balancing change and sustain talk, and eliciting change behavior will all be used accordingly during the sessions. Coaching is tied to the overall results in investigating if motivational interviewing and coaching are effective in increasing movement in populations with cerebral palsy.
  Other Names: Coaching

SUMMARY:
Individuals with cerebral palsy are known to have a reduced amount of physical activity; yet, there are no known intervention strategies for improving the number of steps they take each day. This study will use wearable physical activity monitors to assess if behavioral coaching is a viable strategy for combating the reduced physical activity seen in this patient population.

DETAILED DESCRIPTION:
A lack of physical activity in persons with cerebral palsy is known to have cascading effects on their overall health. Despite this recognition, there have been limited attempts to improve the physical activity of this patient population. The overall landscape of this project is that a cohort of persons with cerebral palsy will undergo 8 weeks of physical activity that is guided by behavioral coaching. This study aims to determine the impact of behavioral coaching on 1) the amount of daily physical activity, 2) changes in the sensorimotor cortical activity, 3) changes in laboratory assessments of functional mobility. The participants with CP will initially undergo neuroimaging and a battery of clinical assessments. After completing the baseline tests, the participants will undergo 8-weeks of behavioral coaching where they are encouraged to increase the number of steps they take per-day. After completing the 8 weeks, the participants will repeat the same assessments that were performed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy diagnosis and ambulatory (Gross Motor Function Classification Score [GMFCS] levels between I-III).

Exclusion Criteria:

* No orthopedic surgery in the last 6 months, botulinum injections within the last 6 months, or metal in their body that would preclude the use of MEG.

Ages: 11 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Mobility Test Time | Baseline and 8 weeks
  The participant will be asked to perform a series of 10-meter walking tasks such as walking at preferred speed, walking as fast as possible, walking while turning the head, walking around cones, and stepping over a box. The participant will also be asked to walk as far as possible for 1 minute. Completion time will be the primary outcome for these tests. Additionally, the tests will also be digitally video-recorded and scored by an independent assessor.
Change in Time in 5 Times Sit-to-Stand | Baseline and 8 weeks
  The participant will start the test by sitting on a bench. The time it takes to stand up and sit down five times will be the outcome measure.
Change in Time for Timed Up and Go | Baseline and 8 weeks
  The participant will start the test by sitting on a bench. The time it takes the participant to stand-up, walk to a line on the floor that is 3-meters away and return to sitting on the bench will be the outcome measure.
Changes in Brain Activity | Baseline and 8 weeks
  Magnetoencephalography (MEG) will be used to assess the changes in the cortical activity while producing a leg motor action and processing peripheral sensations.

CONTACTS AND LOCATIONS:
Locations (1):
- Boys Town National Research Hospital, Boys Town, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI and all of the investigators have made a commitment to publish, in a timely manner, all of the relevant scientific information that they will derive during this project. Deidentified data will be made available upon reasonable request to the Principal Investigator (Dr. Kurz).
Supporting Information: Study Protocol, CSR
Time Frame: Upon completion of study and data analysis
Access Criteria: Contact Dr. Kurz